CLINICAL TRIAL: NCT04521946
Title: A Pilot Study of Allogeneic Hematopoietic Cell Transplantation for Patients With High Grade Central Nervous System Malignancies
Brief Title: Chemotherapy and Donor Stem Transplant for the Treatment of Patients With High Grade Brain Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0495; NCI-2020-05878 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0495 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2023-10

CONDITIONS: Anaplastic Ependymoma; Atypical Teratoid/Rhabdoid Tumor; Central Nervous System Germ Cell Tumor; Choroid Plexus Carcinoma; Intracranial Myeloid Sarcoma; Malignant Brain Neoplasm; Malignant Glioma; Medulloblastoma; Primitive Neuroectodermal Tumor; Recurrent Anaplastic Ependymoma; Recurrent Atypical Teratoid/Rhabdoid Tumor; Recurrent Malignant Brain Neoplasm; Recurrent Malignant Glioma; Recurrent Medulloblastoma; Recurrent Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Ependymoma; Rhabdoid Tumor; Choroid Plexus Carcinoma; Brain Neoplasms; Glioma; Medulloblastoma; Neuroectodermal Tumors, Primitive | interventions — Etoposide; fludarabine phosphate; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation; Antilymphocyte Serum; thymoglobulin; Melphalan; Mycophenolic Acid; Tacrolimus; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, HCT) (Experimental): Patients receive thiotepa IV over 2-4 hours and etoposide IV over 60 minutes on days -8 to -6, melphalan IV over 20 minutes on days -5 and -4, and fludarabine phosphate IV over 1 hour on days -5 to -3. Patients receiving umbilical cord transplant only also receive lapine T-lymphocyte immune globulin IV over 4-12 hours on days -4 and -3. Patients then undergo HCT on day 0. Patients also receive tacrolimus IV or cyclosporine IV beginning on day -2 to and mycophenolate mofetil PO every 8 hours or IV from days 0-40 and tapered to day 90.
  Interventions: Drug: Etoposide; Drug: Fludarabine Phosphate; Procedure: Hematopoietic Cell Transplantation; Biological: Lapine T-Lymphocyte Immune Globulin; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Thiotepa

INTERVENTIONS:
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; Stem Cell Transplant; stem cell transplantation
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-Thymocyte Globulin Rabbit; Grafalon; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; rATG; Thymoglobulin
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO or IV
  Other Names: CellCept; MMF
Drug: Tacrolimus — Given IV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Thiotepa — Given IV
  Other Names: 1,1'',1''''-Phosphinothioylidynetrisaziridine; Girostan; N,N'', N''''-Triethylenethiophosphoramide; Oncotiotepa; STEPA; Tepadina; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312

SUMMARY:
This phase I trial investigates the side effects and effectiveness of chemotherapy followed by a donor (allogeneic) stem cell transplant when given to patients with high grade brain cancer. Chemotherapy drugs, such as fludarabine, thiotepa, etoposide, melphalan, and rabbit anti-thymocyte globulin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving chemotherapy before a donor stem cell transplant helps kill cancer cells in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. When the healthy stem cells from a donor are infused into a patient, they may help the patient's bone marrow make more healthy cells and platelets and may help destroy any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess tolerability of allogenic hematopoietic cell transplantation (HCT) among patients with chemo-responsive high-grade central nervous system (CNS) malignancies as defined by transplant-related mortality (TRM) at day 30 as well as rate of grade III organ toxicity or higher (Bearman Regimen-Related Toxicities Scale) attributable to conditioning occurring within 30 days.

SECONDARY OBJECTIVES:

I. Median time to platelet and neutrophil engraftment. II. Incidence of acute graft-versus-host disease (aGVHD) by day 100. III. Incidence of chronic GVHD at day 100 and one year. IV. Rate of grade II organ toxicity through day 100. V. Rate of graft failure (primary and secondary) through day 100. VI. Rate of infectious complications through day 100. VII. Progression free survival at day 180. VIII. Cumulative incidence of relapse, overall survival, and progression-free survival at 100 days and 1 year.

OUTLINE:

Patients receive thiotepa intravenously (IV) over 2-4 hours and etoposide IV over 60 minutes on days -8 to -6, melphalan IV over 20 minutes on days -5 and -4, and fludarabine phosphate IV over 1 hour on days -5 to -3. Patients receiving umbilical cord transplant only also receive lapine T-lymphocyte immune globulin IV over 4-12 hours on days -4 and -3. Patients then undergo HCT on day 0. Patients also receive tacrolimus IV or cyclosporine IV beginning on day -2 to and mycophenolate mofetil orally (PO) every 8 hours or IV from days 0-40 and tapered to day 90.

After completion of study treatment, patients are followed up at 100, 180, 270 and 360 days.

ELIGIBILITY:
Inclusion Criteria:

* Pathological criteria for any high grade primary or recurrent malignant brain tumor - medulloblastoma (patients who are ineligible for tandem autologous transplants or who are at least 3 months post autologous HCT), primitive neuroectodermal tumor (PNET), atypical teratoid rhabdoid tumor (ATRT), malignant glioma, CNS germ cell tumor, intracranial sarcomas, choroid plexus carcinoma, anaplastic ependymoma. High grade tumors defined as those that are grade III or higher based on World Health Organization (WHO) classification grading system or for medulloblastoma: group 3 and 4 molecular subtypes
* Patients have to be in at least, a chemo-responsive disease status
* Available suitable HCT donor
* Creatinine clearance or glomerular filtration rate (GFR) >= 50 ml/min/1.73m^2, and not requiring dialysis
* Diffusion capacity of the lung for carbon monoxide (DLCO) (corrected for hemoglobin) >= 50% predicted. If unable to perform pulmonary function tests, then O2 saturation >= 92% in room air
* Bilirubin =< 3x upper limit of normal (ULN) (with the exception of isolated hyperbilirubinemia due to Gilbert's syndrome)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 5x for age
* DONOR: HCT will be done using stem cell sources in the following order of preference (and fulfilling minimal cell dose requirements per institutional standards):

  * Matched related donor bone marrow (10 of 10 human leukocyte antigen [HLA] alleles [HLA-A, B, C, DR, and DQ]). Matched related donor peripheral blood stem cell (PBSC) is allowed only if collection of bone marrow (BM) is not available or refused by guardian/donor
  * Matched allogeneic umbilical cord blood: related

    * High-resolution matching at A,B, DRB1 (minimum 4/6)
    * Killer-cell immunoglobulin-like receptor (KIR) major histocompatibility complex (MHC) class 1 preferential mismatch (minimum 4/6)
  * Matched allogeneic umbilical cord blood: unrelated

    * High-resolution matching at A,B, DRB1(minimum 4/6)
    * KIR MHC class 1 preferential mismatch (minimum 4/6)

Exclusion Criteria:

* Lack of histocompatible suitable graft source
* End-organ failure that precludes the ability to tolerate the transplant procedure, including conditioning regimen
* Renal failure requiring dialysis
* Congenital heart disease resulting in congestive heart failure
* Ventilatory failure: requires invasive mechanical ventilation
* Human immunodeficiency virus (HIV) infection
* Uncontrolled bacterial, viral, or fungal infections
* A female of reproductive potential who is pregnant, planning to become pregnant during the study, or is nursing a child
* Any patient who does not fulfill inclusion criteria listed above

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality | At day 30
  Will be reported together with the corresponding 95% Bayesian credible interval. Will be estimated using the method of Gooley.
Rate of grade III or higher organ toxicity attributable to conditioning | Within 30 days
  Assessed per Bearman Regimen-Related Toxicities Scale. Will be reported together with the corresponding 95% Bayesian credible interval.

SECONDARY OUTCOMES:
Failure of platelet and neutrophil engraftment rates | Day 100
  Will be calculated and illustrated from the time of transplant by the method of Kaplan and Meier.
Incidence of acute graft-versus-host (GVHD) disease | Up to day 100
  Will be estimated using the method of Gooley.
Incidence of chronic GVHD | At day 100 and 1 year
  Will be estimated using the method of Gooley.
Rate of grade II organ toxicity | Up to day 100
  Will be reported as counts with percentages.
Rate of graft failure (primary and secondary) | Up to day 100
  Will be reported as counts with percentages.
Rate of infectious complications | Up to day 100
  Will be reported as counts with percentages.
Progression free survival | At day 180
Cumulative incidence of relapse | At day 100 and 1 year
  Will be calculated and illustrated from the time of transplant by the method of Kaplan and Meier.
Overall survival | At day 100 and 1 year
  Will be calculated and illustrated from the time of transplant by the method of Kaplan and Meier.
Progression-free survival | At day 100 and 1 year
  Will be calculated and illustrated from the time of transplant by the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Kris M Mahadeo, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT04521946/ICF_000.pdf